CLINICAL TRIAL: NCT04229030
Title: A Double Blind, Randomized, Multi-Center, Placebo-Controlled Phase 2B Clinical Trial for the Evaluation of Efficacy and Safety of RZL-012 in Subjects Having Dercum's Disease Lipomas
Brief Title: RZL-012 for Dercum's Disease Lipomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RZL-012-DD-P2bUS-001
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2020-01

CONDITIONS: Dercum's Disease Lipomas
MeSH Terms: interventions — RZL-012

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RZL-012 (Active Comparator): A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 4-8 lipomas in each subject, preferably 6. Dosing will be done according to lipomas size, as will be determined by Ultrasound. Each injection contains 0.1mL RZL-012 (5mg).
  Lipomas in the size of:
  2-3.9 cm will be dozed with 0.4mL RZL-012 (20mg). 4-5.9 cm will be dozed with 0.8mL RZL-012 (80mg). 6-7.9 cm will be dozed with 1 mL RZL-012 (100mg). 8-10 cm will be dozed with 1.2 mL RZL-012 (120mg).
  Interventions: Drug: RZL-012
- Vehicle of RZL-012 (Placebo Comparator): A single-treatment injection, multiple subcutaneous injections of vehicle administered into 4-8 lipomas in each subject, preferably 6. Dosing will be done according to lipomas size, as will be determined by Ultrasound. Each injection contains 0.1mL vehicle.
  Lipomas in the size of:
  2-3.9 cm will be dozed with 0.4mL vehicle. 4-5.9 cm will be dozed with 0.8mL vehicle. 6-7.9 cm will be dozed with 1 mL vehicle. 8-10 cm will be dozed with 1.2 mL vehicle.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: RZL-012 — small synthetic molecule for the treatment of Dercum's Disease lipomas
  Arms: RZL-012
Drug: Vehicle — Vehicle of RZL-012 drug product
  Other Names: placebo
  Arms: Vehicle of RZL-012

SUMMARY:
Thirty-eight (38) subjects will be included in the study. Subjects will be randomized in a ration of 1:1 to be treated with RZL-012 or placebo. Subjects will be injected with a different doses of RZL-012 according to their lipomas sizes. The total of 38 subjects will be enrolled in 3 clinical sites.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blind, placebo controlled clinical trial in DD subjects having lipomas. Subjects will be randomized, in a 1:1 ratio, into two groups injected with either RZL-012 or vehicle.

Once the study ends and codes are opened, 84 days after dosing, placebo-treated subjects will be offered the option of receiving treatment with RZL-012 and followed up for an additional 84 days.

At least 4 lipomas/nodules, preferably 6, and no more than 8, will be injected per subject, two of which will be medium (4-5.9 cm), large (6-7.9 cm) or extra-large (8-10 cm) in diameter. Dosing will be according to lipoma size, where the total injected dose will not exceed 240 mg per patient (48 injections at 5mg/injection).

ELIGIBILITY:
Inclusion Criteria:

* At least 4 painful lipomas of appropriate size to be injected on a background of Dercum's Disease.
* Generally considered healthy according to medical history, physical examination, electrocardiogram (ECG) and laboratory evaluation with an emphasis on metabolic parameters (fasting glucose concentration < 200 mg/dL).
* Subjects must be able to adhere to the visit schedule and protocol requirements and be capable of completing the study.
* Males or females in the age of fertility are willing to refrain from sexual activity or agree to use a double-barrier contraceptive device (e.g., condom and spermicide) for 4 weeks after treatment with RZL 012.
* Subjects must sign an informed consent indicating they are aware of the investigational nature of the study.

Exclusion Criteria:

* Unable to tolerate subcutaneous injections.
* Pregnant women.
* Subjects with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorders, that in the opinion of the investigator places the subject at significant risk.
* Positive blood screen for Hepatitis B surface antigen (HbSAg), Hepatitis C virus (HCV), or Human immunodeficiency virus (HIV).
* Subjects with a clinical history of active primary or secondary immunodeficiency, autoimmune disease or subjects taking immunosuppressive drugs such as corticosteroids
* Subjects with dysfunctional gallbladder activity, e.g. underwent cholecystectomy or cholecystitis.
* As a result of medical review and physical examination, the PI (or medically qualified nominee) considers the subject unfit for the study.
* Known sensitivity to components of the injection formulation.
* Prior wound, tattoo or infection in the treated area.
* Prior invasive treatment such as surgery or injectable drug at the RZL-012 injected area.
* Subjects treated chronically at least 3 months prior to study entry with systemic steroids or immunosuppressive drugs.
* Subjects treated chronically at least one week prior to study entry with Non-Steroidal Anti-Inflammatory Drugs (NSAIDs).
* Current participation or participation within 3 months prior to the start of this study in a drug or other investigational research study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Limitless Therapeutics, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: lipomas
Groups:
- RZL-012: A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 4-8 lipomas in each subject, preferably 6. Dosing will be done according to lipomas size, as will be determined by Ultrasound. Each injection contains 0.1mL RZL-012 (5mg).
  Lipomas in the size of:
  2-3.9 cm will be dozed with 0.4mL RZL-012 (20mg). 4-5.9 cm will be dozed with 0.8mL RZL-012 (80mg). 6-7.9 cm will be dozed with 1 mL RZL-012 (100mg). 8-10 cm will be dozed with 1.2 mL RZL-012 (120mg).
  RZL-012: small synthetic molecule for the treatment of Dercum's Disease lipomas
- Vehicle of RZL-012: A single-treatment injection, multiple subcutaneous injections of vehicle administered into 4-8 lipomas in each subject, preferably 6. Dosing will be done according to lipomas size, as will be determined by Ultrasound. Each injection contains 0.1mL vehicle.
  Lipomas in the size of:
  2-3.9 cm will be dozed with 0.4mL vehicle. 4-5.9 cm will be dozed with 0.8mL vehicle. 6-7.9 cm will be dozed with 1 mL vehicle. 8-10 cm will be dozed with 1.2 mL vehicle.
  Vehicle: Vehicle of RZL-012 drug product
Period: Overall Study
Arm/Group | RZL-012 | Vehicle of RZL-012
Started | 20; 125 lipomas | 18; 109 lipomas
Completed | 20; 125 lipomas | 18; 109 lipomas
Not Completed | 0; 0 lipomas | 0; 0 lipomas

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RZL-012 | Vehicle of RZL-012 | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.4) | 48 (12.4) | 50.15 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Change in Lipomas Dimensions
Description: Evaluation of the efficacy of RZL-012 following injection into lipomas/nodules of Dercum's Disease (DD) subjects. Efficacy will be determined by ultrasound assessment of the lipoma/nodule dimensions after treatment vs baseline. Lipomas Dimensions will be measured for active vs. placebo at days 28,56,84
Time Frame: 0-84 days
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | RZL-012 | Vehicle of RZL-012
Number analyzed (Participants) | 20 | 18
percentage of change from baseline | -15.13 (25.56) | -15.92 (23.96)

2. Secondary Outcome: Key Secondary Outcome - Efficacy - Improvement in Pain Assessment of Individual Lipomas
Description: Assessment of lipoma/nodule associated pain using the Comparative Pain Scale. 0 is "no pain" and 10 is "worst pain". Pain measured for active vs. placebo at days 28,56,84
Time Frame: 0-84 days
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | RZL-012 | Vehicle of RZL-012
Number analyzed (Participants) | 20 | 18
percentage of change from baseline | -56.15 (35.77) | -34.34 (40.15)

3. Secondary Outcome: Safety Number of Participants With One or More Abnormal Laboratory Values up to Day 28
Description: Safety will be assessed by by change-from-baseline values for clinical laboratory tests. measured for active vs. placebo at days 1 and 28 following injection. Number of subjects with abnormal laboratory values will be compared in both study arms.
Time Frame: 0-28 days
Measure: Count of Participants; unit: Participants
Arm/Group | RZL-012 | Vehicle of RZL-012
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

4. Other Pre Specified Outcome: Exploratory
Description: Improvement in Quality of Life - QOL questionnaire. Improvement will be measured for active vs. placebo at Day 0 and Day 84 following treatment.
Time Frame: 0-84 Days
Measure: Count of Participants; unit: Participants
Arm/Group | RZL-012 | Vehicle of RZL-012
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | RZL-012 | Vehicle of RZL-012
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 20/20 | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RZL-012 (N=20) | Vehicle of RZL-012 (N=18)
Injection site bruising (General disorders) | 6 | 3
Injection site discoloration (General disorders) | 5 | 0
Injection site erythema (General disorders) | 20 | 17
Injection site hypesthesia (General disorders) | 2 | 0
Injection site edema (General disorders) | 20 | 18
Injection site pain (General disorders) | 11 | 9
Injection site pruritus (General disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT04229030/Prot_SAP_000.pdf